CLINICAL TRIAL: NCT00247013
Title: Automated Tele Counseling for Screening Mammography
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: R01CA084447-01 (NIH); National Cancer Institute
Record Dates: First submitted 2005-10-28; First posted 2005-11-01 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2010-09

CONDITIONS: Breast Cancer
Keywords: automated telephone system; breast cancer; cancer prevention; intervention; mammography; screening
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Behavioral: Breast Cancer Screening Compliance

SUMMARY:
The purpose and aim of this study is to test the use of a computer-based, automated telecommunications system and its effectiveness in increasing the rates of regular screening mammography among women ages 50-74. The system will not only help in scheduling appointments but will help women in overcoming any barriers that may deter them from having the procedure at all. The programs are designed to be user friendly and easy to implement in clinical practice.

DETAILED DESCRIPTION:
The primary goal of this project is to evaluate the effectiveness and acceptability of a computer-based telecommunications system for increasing rates of regular screening mammography among women ages 50-74. The Telephone-Linked-Communications for Mammography Screening (TLC-M) is designed to educate, advise and motivate women to have regular screening mammograms. There will be two versions of TLC-M: one for women who are coming due for their annual screening mammography ("pre-due" women) and one for women who have missed their annual mammogram ("past-due" women). TLC-M uses a real human voice to speak to the women on the telephone; the subjects communicate by using the touch tone keypad on their telephones. The intervention will consist of up to three automated telephone conversations. During the call TLC-M assesses the woman's willingness to have a mammogram, helps interested women schedule a mammogram, and identifies and addresses difficulties or barriers she might have in getting a mammogram. This study will consist of two linked randomized controlled trials. We will recruit 2,120 participants over 12 months from two radiology departments. Three to four months prior to their due date for an annual screening mammogram, these women will receive a reminder letter to schedule a mammogram. In addition, a random sample of them will use TLC-M. All participants in this "pre-due" intervention study will be evaluated 3 months after their due date to determine whether or not they obtained a mammogram. Of the women who received the letter only in the first trial, those who did not obtain a mammogram during the observation period will enter a "past due" intervention trial. These women will be randomly assigned to receive a "past due" reminder letter or to use the TLC-M. Four months later, participants will be evaluated to determine whether they had a mammogram. For both trials mammography rates of those women who used the TLC-M and those who did not will be statistically compared.

ELIGIBILITY:
Inclusion Criteria:

* Ages 50-74
* A recent (within the last 6 months) negative screening mammogram

Exclusion Criteria:

* Lack a permanent address or planning to move from the Boston area during the study period
* No home telephone or no touch tone service
* Cannot use a telephone unassisted
* Cannot understand conversational English over the telephone
* Major medical illness that would preclude participation
* History of breast cancer
* Mammography or other breast diagnostic procedures (except CBE) or therapeutic procedures since the last screening mammogram
* Another member of household enrolled in the study (to eliminate possible study contamination)

Ages: 50 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2120
Dates: Start 1996-01; Study Completion 2006-01

PRIMARY OUTCOMES:
Number of women who have repeat screening mammogram

SECONDARY OUTCOMES:
Evaluation of intervention for those women who used TLC-M

CONTACTS AND LOCATIONS:
Overall Officials: Robert Friedman, MD, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States